CLINICAL TRIAL: NCT02749331
Title: Study of Recombinant Adenovirus (AdVince) in Patients With Neuroendocrine Tumors; Safety and Efficacy
Brief Title: Study of Recombinant Adenovirus AdVince in Patients With Neuroendocrine Tumors; Safety and Efficacy
Acronym: RADNET
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Uppsala University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VIRUSNET201401; 2014-000614-64 (EudraCT Number)
Record Dates: First submitted 2016-03-11; First posted 2016-04-22 (Estimated); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Neuroendocrine Tumors
MeSH Terms: conditions — Neuroendocrine Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- AdVince (Experimental): Dose escalation, minimum 3 patients per dose in Phase I. Dose levels:
  1. 10 000 000 000 virus particles
  2. 100 000 000 000 virus particles
  3. 300 000 000 000 virus particles
  4. 1000 000 000 000 virus particles
  Maximum tolerated dose will be confirmed by 12 additional patients treated at this dose level in Phase IIa.
  Interventions: Drug: AdVince

INTERVENTIONS:
Drug: AdVince — Virus solution for infusion in intrahepatic artery
  Other Names: Ad5PeptideTransductionDomain(PTD)(CgA-E1AmiR122)

SUMMARY:
An open-labelled, uncontrolled, single-center Phase I/IIa clinical study to evaluate the safety of repeated infusions of AdVince into the hepatic artery in patients with metastatic neuroendocrine tumors (NETs), and if possible determination of maximum tolerated dose.

DETAILED DESCRIPTION:
An open-labelled, uncontrolled, single-center Phase I/IIa clinical study to evaluate the safety of repeated infusions of AdVince into the hepatic artery in patients with metastatic neuroendocrine tumors (NETs), and if possible determination of maximum tolerated dose. Secondary objectives include to evaluate the anti-tumoral efficacy of AdVince infusions on metastatic neuroendocrine tumors, to determine the replication profile of AdVince and to determine the humoral (antibody) and cytokine-mediated immune response to AdVince. Minimum 12 and maximum 35 patients will be included, the number is based on the toxicity observed.

ELIGIBILITY:
Inclusion Criteria:

1. Subject´s written informed consent
2. Histologically and radiologically confirmed progressive neuroendocrine carcinoma of gastrointestinal, pancreatic or bronchial origin with multiple liver metastases. Progression in Clinical symptoms and tumor growth verified over the last 6 months on CT or MRI
3. Cancer that is not considered resectable for potential cure or tumor reduction
4. Patent portal vein and adequate liver perfusion
5. Liver dominant disease with involvement of <60% of liver parenchyma
6. Karnofsky performance status of >=70%
7. Life expectancy of >=6 months
8. >=18 years of age
9. Must use a reliable method of contraception if sexually active and of reproductive potential
10. Plasma creatinine <105 ug/ml
11. Aspartate transaminase (AST), Alanine transaminase (ALT) and Alkaline Phosphatase (ALP) <3.0-fold upper limit of normal
12. Total bilirubin <2.0-fold upper limit of normal
13. Prothrombin time (PT)/International Normalized Ratio (INR) <2.0 and Prothromboplastin time (PTT) within normal limits
14. Neutrophils >1500/ml, hemoglobin >100 g/L, platelets >100 000/ml
15. Patients with functioning NET should have cover by somatostatin analog

Exclusion Criteria:

1. Known chronic liver dysfunction Before the development of metastatic cancer (e.g. cirrhosis, chronic hepatitis)
2. Active infection, including documented HIV and hepatitis C
3. Any viral syndrome diagnosed within the previous 2 weeks
4. Chemotherapy within the previous 4 weeks Before the first treatment
5. Radiotherapy to the target tumor site within the last 24 weeks from the baseline CT scan
6. Concomitant malignancy
7. Pregnant or lactating females
8. Prior participation in any research protocol that involved administration of adenovirus vectors
9. Treatment with any other investigational therapy within the last 4 weeks, organ transplantation prior to treatment, severe cardiovascular, metabolic or pulmonary disease
10. Continuing treatment with any other cancer therapy

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2016-03 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Number of Adverse Events (AE) according to Common Terminology Criteria for Adverse Events (CTCAE) v 4.03 | From screening visit and through study completion, an average time of 18 months.
  AEs probably or possibly related to the study drug or local injuries caused by the administration procedure. If possible identify dose limiting toxicity (DLT), i.e. grade 4 toxicity of any duration or grade 3 toxicity lasting more than 7 days, excluding flu-like symptoms, according to CTCAE v4.03.Clinically significant changes in laboratory parameters (haematology, blood coagulation, liver function, biochemistry and kidney function) and vital signs (body temperature, heart rate, blood pressure, respiratory rate and consciousness according to Reaction Level Scale from 1985 (RLS-85).

SECONDARY OUTCOMES:
Change in tumor size | Measured within 4 weeks before first treatment and after 80 +/-14 days (evaluation visit 1)
  Computer tomography (CT) and/or positron emission tomography (PET) with magnetic resonance imaging (MRI). Assessment based on Response Evaluation Criteria In Solid Tumors (RECIST) or modified RECIST (mRECIST).
Change in tumor size | Measured within 4 weeks before first treatment and after 214 +/- 14 days (evaluation visit 2)
  Computer tomography (CT) and/or positron emission tomography (PET) with magnetic resonance imaging (MRI). Assessment based on Response Evaluation Criteria In Solid Tumors (RECIST) or modified RECIST (mRECIST).
Change in tumor metabolic activity | Baseline value within 24 hrs before first treatment and after 80 +/- 14 days(evaluation visit 1)
  Change in hormone levels including chromogranin- A (CgA), chromogranin-B (CgB), neuron specific enolase (NSE) and specific hormones.
Change in tumor metabolic activity | Baseline value within 24 hrs before first treatment and after 214 +/- 14 days (evaluation visit 2)
  Change in hormone levels including chromogranin- A (CgA), chromogranin-B (CgB), neuron specific enolase (NSE) and specific hormones.
Progression-free survival (PFS) | Twelve weeks after 80 days from first treatment (4 treatment cycles) or the corresponding time.
  Number of patients with progression-free survival (PFS).
Change in replication profile of AdVince | Before and 4hrs after each treatment cycle up to a time period of 214 days.
  Replication profile determined by quantification of adenovirus genomic copies in patient´s blood by quantitative real-time polymerase chain reaction (QRT-PCR).
Change in replication profile of AdVince | Before and 24hrs after each treatment up to a time period of 214 days.
  Replication profile determined by quantification of adenovirus genomic copies in patient´s blood by quantitative real-time polymerase chain reaction (QRT-PCR).
Change in replication profile of AdVince | Before and 72hrs after each treatment cycle up to a time period of 214 days.
  Replication profile determined by quantification of adenovirus genomic copies in patient´s blood by quantitative real-time polymerase chain reaction (QRT-PCR).
Change in the humoral immune response to AdVince | At baseline, after 8+2 days, after 50 +/- 7days, optional after 124 +/- 7days and 184 +/- 7 days.
  Detection of anti-adenovirus neutralizing antibodies against adenovirus.
Change in the cytokine-mediated immune response | At baseline and at 4hrs following each treatment up to a time period of 214 days.
  Measure from patient´s plasma.
Change in the cytokine-mediated immune response | At baseline and at 24hrs following each treatment up to a time period of 214 days.
  Measure from patient´s plasma.
Change in the cytokine-mediated immune response | At baseline and at 72hrs following each treatment up to a time period of 214 days.
  Measured from patient´s plasma.

CONTACTS AND LOCATIONS:
Overall Officials: Joakim Crona, MD, PhD, Principal Investigator — Uppsala University Hospital
Locations (1):
- Endocrine Oncology Clinic, Uppsala University Hospital, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: No